CLINICAL TRIAL: NCT06120985
Title: Expanding Safe Water Access to Improve Health Outcomes in Rural Appalachia: A Pilot Water Treatment Intervention Trial in Virginia & Tennessee
Brief Title: Rural Appalachia Pilot Water Treatment Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: East Tennessee State University (Other); University of North Carolina, Chapel Hill (Other); Ballad Health (Other)
Responsible Party: Principal Investigator, Alasdair Cohen, Assistant Professor of Environmental Epidemiology, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-685
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Water-Related Diseases; Enteric Pathogens; Exposure to Chemical Pollution
MeSH Terms: conditions — Waterborne Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Households randomized to the treatment group will be provided countertop pitcher water filters
  Interventions: Device: Countertop pitcher water filter
- Control (No Intervention): Households randomized to the control group will be provided water filters at the completion of the study

INTERVENTIONS:
Device: Countertop pitcher water filter — Point-of-use drinking water filter
  Arms: Treatment

SUMMARY:
Consumption of unsafe drinking water is associated with a substantial burden of disease globally. In the USA, the burden of disease associated with consumption of contaminated drinking water from non-regulated private wells and springs in rural areas is relatively understudied and unclear. For some lower-income households in rural areas of the USA without access to reliably safe drinking water, point-of-use treatment with relatively low-cost pitcher filters could help to reduce exposures to contaminated water and associated adverse health outcomes. This pilot randomized controlled intervention trial will provide information and data on water quality and contamination exposures, associated health outcomes, and the adoption potential of point-of-use water filters in rural areas of Virginia and Tennessee.

ELIGIBILITY:
Inclusion Criteria:

* The household does not have utility-supplied water at the time of enrollment,
* The household is considered to be "low-income" (based on federally defined income limits),
* The household is in one of the selected study counties in TN or VA.

Exclusion Criteria:

* None (no exclusion criterion based on gender, race, ethnicity, language, or literacy).

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
E. coli detection in drinking water | 12 months
  Proportion of households with E. coli (indicator of fecal contamination) detected in drinking water samples
Heavy metals or other contaminants exceeding EPA MCL | 12 months
  Proportion of households with contaminants detected in drinking water at concentrations exceeding the US Environmental Protection Agency (EPA) Safe Drinking Water Act (SDWA) Maximum Contaminant Levels (MCL)

SECONDARY OUTCOMES:
Gastrointestinal illness | 12 months
  Incidence of acute gastrointestinal illness via self-reported diarrhea (7-day recall)
Pathogen infection | 12 months
  Detection of enteric pathogen infection via qPCR analysis of stool samples and salivary antibody assays

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Cohen, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - East Tennessee State University, Johnson City, Tennessee
  - Virginia Tech, Blacksburg, Virginia